CLINICAL TRIAL: NCT03772938
Title: Stem Cells Therapy in Degenerative Diseases of the Retina
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Marta P. Wiącek, MD, PhD candidate, principal investigator, Pomeranian Medical University Szczecin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IKiKO-KB-0012/143/13
Record Dates: First submitted 2018-11-03; First posted 2018-12-12 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Retinal Degeneration; Retinitis Pigmentosa; Age Related Macular Degeneration; Stargardt Disease 1
Keywords: stem cells; Retinitis Pigmentosa; Age Related Macular Degeneration; Stargardt Disease; electroretinography
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Macular Degeneration; Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem/progenitor cells transplantation (Active Comparator): Intervention: A single intravitreal injection of autologous bone marrow-derived stem/progenitor cells will be performed.
  Interventions: Biological: Stem/progenitor cells transplantation
- Standard treatment of degenerative disease of retina (Sham Comparator): Symptomatic treatment of degenerative disease of retina without biologic cell-based treatment
  Interventions: Biological: Stem/progenitor cells transplantation

INTERVENTIONS:
Biological: Stem/progenitor cells transplantation — Human autologous bone marrow-derived stem/progenitor cell transplantation administered as an intravitreal injection in patients with degenerative disease of retina.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an autologous bone marrow-derived stem/progenitor cells administered intravitreously in the subjects with degenerative diseases of the retina.

DETAILED DESCRIPTION:
Degenerative diseases of the retina are challenging for ophthalmologists. This is a common term that covers heterogenous group of diseases, f.e. retinitis pigmentosa, Stargardt disease, Best's disease or age related macular degeneration. Undetermined etiology, wide range of factors that may trigger the onset of the disease and modulate it's course impede the implementation of an effective treatment. Currently, a stem cells therapy seems to be promising option in patients with degenerative diseases of the retina. The purpose of this prospective, nonrandomized, open label, pilot study is to conduct the investigation of the safety and efficacy of intravitreal injection of autologous bone marrow-isolated stem/progenitor cells with different selected phenotypes into the subjects with degenerative diseases of the retina. Especially, this clinical trial is designated to test the therapeutic (pro-regenerative and neuro-protective) functions of different stem/progenitor cell populations able to secrete bioactive neurotrophic factors. All patients enrolled will have a documented history of degenerative disease of the retina prior to study enrollment. Next, autologous bone marrow-isolated stem/progenitor cells intravitreous injection will be performed. Finally, treatment safety, adverse events and exploratory parameters, including best corrected visual acuity, visual field and electroretinography parameters, to establish disease progression rate will be recorded throughout the duration of the post-treatment follow up period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed degenerative disease of the retina,
* age 18-65 years,
* best corrected visual acuity max. 0,2 (Snellen letter chart),
* good understanding of the protocol and willingness to consent,
* signed informed consent.

Exclusion Criteria:

* concomitant eye disease (glaucoma, etc.)
* concomitant of other systemic disease or diseases,
* inflammation (high protein or lymphocytosis in the CSF), active infections.
* diabetes,
* cardio-vascular disorders,
* cancer,
* autoimmune diseases,
* renal failure,
* impaired hepatic function,
* subject unwilling or unable to comply with the requirements of the protocol,
* patient has been treated previously with any cellular therapy,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  Confirm the safety of autologous bone marrow stem/progenitor cell intravitreal injection in enrolled patients by repeated follow-up over one year with clinical evaluations.

SECONDARY OUTCOMES:
Efficacy of autologous bone marrow stem/progenitor intravitreal injection in enrolled patients. | 12 months
  Best corrected visual acuity, ETDRS chart [number of letters]
Intraocular pressure | 12 months
  Pascal tonometer [mmHg]
Optic disk retinal nerve fiber layer | 12 months
  optical coherence tomography [um]
Central macular thickness | 12 months
  optical coherence tomography [um]
Ganglion cell complex thickness | 12 months
  optical coherence tomography [um]
Choroidal thickness | 12 months
  Enhanced depth imaging optical coherence tomography [um]
Choroidal volume | 12 months
  Enhanced depth imaging optical coherence tomography [mm3]
Computed perimetry (30-2 and 10-2 module) | 12 months
  mean deviation, pattern standard deviation [B]
Goldmann perimetry with color filters | 12 months
  [degrees]
Contrast sensitivity | 12 months
  Pelli-Robson chart [number of letters]
Function of the photoreceptors (rods and cones), inner retinal cells (bipolar and amacrine cells), and ganglion cells. | 12 months
  Electroretinography (ERG) examination:
  * amplitude of a and b waves [V],
  * culmination time of a and b waves [s],
  * culmination time of q1-q3 waves [s].
Function of the photoreceptors | 12 months
  Multifocal electroretinography (mfERG) examination:
  * retinal response density [V/degree 2],
  * culmination time of P1 wave in 6 rings [s].
Function of ganglion cells | 12 months
  Pattern electroretinography (PERG) examination:
  * amplitude of P50 and N95 waves [V],
  * culmination time of P50 wave [s].

CONTACTS AND LOCATIONS:
Overall Officials: Bogusław Machaliński, MD, PhD, Study Chair — Pomeranian Medical University; Anna Machalińska, MD, PhD, Study Director — Pomeranian Medical University
Locations (1):
- I Department of Ophthalmology, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No